CLINICAL TRIAL: NCT05919589
Title: Evaluating Care Integration for Children with Special Health Care Needs
Brief Title: Evaluating Care Integration for Children with Special Health Care Needs V1.0
Status: Recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: IRAS - 317445
Record Dates: First submitted 2023-06-09; First posted 2023-06-26 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-03

CONDITIONS: Parents; Staff Attitude; Healthy
Keywords: Children with special healthcare needs; CSHCN; Parents; Carer; Professionals; Staff

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Parents and Carers: Parents and carers of children with special healthcare needs
  Interventions: Other: Care Integration for Children With Special Health Care Needs
- Staff and professionals: Staff and professionals involved (either directly or indirectly in healthcare and other services) with children with special healthcare needs
  Interventions: Other: Care Integration for Children With Special Health Care Needs

INTERVENTIONS:
Other: Care Integration for Children With Special Health Care Needs — The Evelina London Children's Hospital (ELCH) is planning to integrate care for children with special health care needs (CSHCN) using a package of support, including 1) family support workers to manage care coordination and support parents, and 2) 'navigation' packs outlining key services, for both the services users and providers

SUMMARY:
The Evelina London Children's Hospital (ELCH) is planning to integrate care for children with special health care needs (CSHCN) using a package of support, including 1) family support workers to manage care coordination and support parents, and 2) 'navigation' packs outlining key services, for both the services users and providers.

This study aims to explore the views and experiences of key stakeholders involved with these services, including the parents/caregivers of CSHCN, and professionals/staff team members. These will be explored using semi-structured qualitative interviews.

DETAILED DESCRIPTION:
There has been a push at the policy level to implement integrated care approaches in the USA and the UK. However, few integrated care models have been evaluated, particularly for children with special health care needs (CSHCN). This is an important group with high levels of needs, and complex and intensive use of services, and which the research team hypothesize could benefit immensely from care integration. This project aims to qualitatively evaluate care integration implementation for CSHCN, to understand how and why integrated services do (or do not) work to improve integration of care.

This research gap was confirmed by a systematic literature review on these topics, conducted by the research team (in final draft stages). The research team also facilitated workshops with local families of CSHCN and professionals to understand their experiences of care delivery, current concerns, and what should be improved.

Synthesizing information from both the systematic literature review and the workshops led to the development of this research project, which will investigate how care can be better integrated for CSHCN and their families.

The themes to be investigated will include:

i. To explore the perceptions of key stakeholders on the overall quality of life, wellbeing, and community inclusion of CSHCN and their parents/caregivers.

ii. To explore the perceptions of key stakeholders on CSHCN and family satisfaction with care, and care integration, including equity of access and how this is impacted by integration.

iii. To explore the views of key stakeholders on the impact of the new key worker/care-coordinator service on the CSHCN and family, including school, work, family, and healthcare use.

With the learning from this project, the research team also aim to develop a model of care that can be evaluated at a larger scale in a later study and, if shown to be successful, delivered throughout the NHS and internationally.

ELIGIBILITY:
Inclusion Criteria:

* Parents/care givers of CSHCN
* Staff and professional stakeholders involved (either directly or indirectly) with CSHCN

Exclusion Criteria:

* Participants under the age of 18 years
* Participants who are unable to speak and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parents/carers of children with special health care needs (CSHCN) attending/referred to paediatric settings of Evelina London Children's Hospital (ELCH), clinical care team members from the paediatrics settings of ELCH, commissioners from Lambeth and Southwark, community health team involving CSHCN in Lambeth and Southwark, and other key stakeholders from the local NHS trust and other organisations
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in perceptions of care integration for children with special healthcare needs (CSHCN) identified though qualitative interviews from baseline to follow-up | Baseline at the start of the intervention, and follow-up after at least 1 month of the intervention.
  Exploring views and experiences of participants on how can care be better integrated for children with special healthcare needs (CSHCN), and their families using a 'Topic guide' through a semi-structured qualitative interview. The topic guide was developed based on present available literature on the role of a care coordinator for CSHCN and discussions with families, colleagues from paediatrics clinical team at ELCH, and the community health team for Lambeth and Southwark.

CONTACTS AND LOCATIONS:
Locations (1):
- St Thomas' Hospital, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goodwin N. Understanding Integrated Care. Int J Integr Care. 2016 Oct 28;16(4):6. doi: 10.5334/ijic.2530. No abstract available. PMID 28316546
- See also: Report to Congress: National Strategy for Quality Improvement in Health Care. March 2011. Submitted by the U.S. Department of Health and Human Services. — http://archive.ahrq.gov/workingforquality/reports/2011-annual-report.html
- See also: Integrated Care: Our Shared Commitment. A framework that outlines ways to improve health and social care integration. From: Department of Health & Social Care — http://assets.publishing.service.gov.uk/government/uploads/system/uploads/attachment_data/file/198748/DEFINITIVE_FINAL_VERSION_Integrated_Care_and_Support_-_Our_Shared_Commitment_2013-05-13.pdf